CLINICAL TRIAL: NCT05187247
Title: Virtual Reality Glasses During Extra-Amniotic Balloon Insertion for Pain and Anxiety Relieve - a Randomized Controlled Trial
Brief Title: VR Glasses During Induction of Labour for Pain and Anxiety Relieve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, ilia kleiner, Obstetrics and Gynecology Resident, MD, Principal investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0156-21-WOMC
Record Dates: First submitted 2021-11-23; First posted 2022-01-11 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Virtual Reality; Induction of Labor Affected Fetus / Newborn; Extra Amniotic Balloon
Keywords: Virtual reality; Induction of Labor; Extra amniotic Balloon

STUDY DESIGN:
Intervention Model Description: A pregnant women who is designated for induction of labor using an extra-amniotic balloon catheter will complete a STAI questionnaire about the degree of anxiety prior to the procedure. All women then will be randomly assigned to 2 groups according to a randomization table. Women assigned to the VR group will use the "virtual reality" technology throughout the insertion procedure while the second group will constitute a control group for the intervention group.
  During the insertion procedure, a subjective assessment of the degree of pain will be performed using VAS score (Visual Analog Scale), and objective pain assessment which will be performed by measuring a pulse at a predetermined time points.
  At the end of the procedure the women will be asked to answer another anxiety questionnaire.
  Women in the VR group will also answer a satisfaction questionnaire from the experience
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Women assigned to the VR group will use the "virtual reality" technology throughout the insertion procedure
  Interventions: Device: Virtual Reality glasses
- control group (No Intervention): control group for the intervention group

INTERVENTIONS:
Device: Virtual Reality glasses — use of virtual reality glasses to reduce anxiety and pain levels
  Arms: VR group

SUMMARY:
In the current study, The investigators aim is to test the distraction affect of "Virtual Reality" (VR) technology on pain and anxiety in pregnant women who undergo through an induction of labour with an extra-amniotic balloon catheter

DETAILED DESCRIPTION:
Insertion of Extra-Amniotic Balloon (EAB) is a recommend mechanical method of Induction of labour. This method of induction causes the cervix to dilate through mechanical pressure on the cervix.

During the procedure of insertion the women is lying on her back. Insertion of EAB is performed by conventional means.

The insertion of EAB can involve discomfort, pain and anxiety before and during the procedure.

While there are numerous studies which describe interventional, pharmacological and non-pharmacological means for pain and anxiety relieve during latent and active phase of labour, there is no sufficient evidence for pain and anxiety relieve during the pre-labour and through induction of labour period.

The "Virtual Reality" (VR) technology is a simple non-invasive technology. The advantage of VR is that it can distract the patient's attention from pain and anxiety by exposure to a virtual reality environment. This technology uses processes of sight, and hearing that requires attention.

Many studies have already investigated the use of VR technology in various medical procedures, such as dental treatment, infusion, pediatric treatment, burns, trauma, chemotherapy, diagnostic hysteroscopies and other medical procedures that are common to the patient's experience of pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women going through mechanical induction of labour with Extra-Amniotic Balloon

Exclusion Criteria:

* Women with history of migraine, headache, epilepsy, vestibular disorders
* Women suffering from seasickness ,motion sickness, vertigo, nausea, vomiting, seizures

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 145 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity | 1 hour
  Subjective assessment of the degree of pain would be graded according to the VAS (Visual Analogue Scale) which is a scale used to measure subjective pain intensity according to a pain scale of 0 to 10, An objective pain assessment will be performed by measuring a pulse at a predetermined time points.

SECONDARY OUTCOMES:
Change in Anxiety state | 1 hour
  Anxiety levels will be measured by a valid questionnaire for assessing situational anxiety called The State-Trait Anxiety Inventory (STAI: Y). This version includes 20 statements which represents feelings that characterize anxiety. Women will be asked to rate them on a scale between 1 to 4. The final score in each questionnaire is obtained by summarizing all the ratings. A higher score indicates a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: ilia kleiner, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Lim SE, Tan TL, Ng GYH, Tagore S, Kyaw EEP, Yeo GSH. Patient satisfaction with the cervical ripening balloon as a method for induction of labour: a randomised controlled trial. Singapore Med J. 2018 Aug;59(8):419-424. doi: 10.11622/smedj.2018097. PMID 30175373
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Derived] Kleiner I, Mor L, Friedman M, Abeid AA, Shoshan NB, Toledano E, Bar J, Weiner E, Barda G. The use of virtual reality during extra-amniotic balloon insertion for pain and anxiety relief-a randomized controlled trial. Am J Obstet Gynecol MFM. 2024 Jan;6(1):101222. doi: 10.1016/j.ajogmf.2023.101222. Epub 2023 Nov 10. PMID 37951577